CLINICAL TRIAL: NCT02483130
Title: A Randomised Controlled Double Blind Crossover Study of the Effect of a Single Dose of N-acetylcysteine Versus Placebo on Brain Glutamate in Patients With Psychotic Disorders
Brief Title: Effect of N-acetylcysteine on Brain Glutamate
Acronym: NAC
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: BRCNAC
Record Dates: First submitted 2015-06-24; First posted 2015-06-26 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2016-08

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders | interventions — Acetylcysteine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples are collected for two purposes.
  1. Participants are invited to donate samples to the BRC Bioresource. These samples may be used in the future for genetic, epigenetic, metabolomic or proteomic analysis.
  2. Participants will also be asked for a blood sample after completion of each MRI scan. These will be used to measure blood glutathione levels, which may be altered by N-acetylcysteine and therefore provide indication of pharmacological effect.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NAC or Placebo: Participants will receive 2400mg capsules of N-Acetylcysteine or placebo
  Interventions: Dietary Supplement: N-Acetylcysteine; Other: Placebo

INTERVENTIONS:
Dietary Supplement: N-Acetylcysteine — Participants will receive 2400mg of N-Acetylcysteine orally via 6 x 400mg capsules.
Other: Placebo — Participants will receive 2400mg of placebo orally via 6 x 400mg capsules.

SUMMARY:
A double-blind, placebo controlled, crossover study to determine whether a single dose of N-acetylcysteine (a nutritional supplement) can reduce brain glutamate levels in patients with a psychotic disorder. Secondary outcomes are to determine the pattern of alteration in brain perfusion and activity following a single dose of N-acetylcysteine.

DETAILED DESCRIPTION:
This is a physiological, proof-of-concept study designed to investigate whether a single administration of N-acetylcysteine can reduce brain glutamate levels in people with psychotic disorders.

Previous research suggests that poor response to antipsychotics may be linked to increased levels of glutamate in the brain (Egerton et al., 2012; Demjaha, Egerton et al., 2013). Reducing brain glutamate levels may therefore be therapeutic. This study tests whether it is possible to reduce brain glutamate levels in psychotic disorders.

This is a small pilot study to determine whether a single administration of NAC can reduce brain glutamate levels in psychosis. At the same time, we will also examine the effects of NAC on brain resting perfusion and activity, to gain more information about how NAC may be acting.

This study will recruit participants with a previous diagnosis of a psychotic disorder. There will be three study visits, 1-2 weeks apart. The first visit will involve a physical health check, blood sample and an interview to assess current symptoms and confirm medical history. On the second and third visits participants will have an MRI scan, lasting one hour, after taking capsules containing either 2400mg NAC or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Diagnosis of a psychotic disorder
* Have mental capacity to consent

Exclusion Criteria:

* Diagnosed drug or alcohol dependency, with the exception of nicotine
* Pregnancy, as determined through a urine pregnancy test
* Presence of any physical health abnormality which may impact on safety to participate in the research, as determined by a study clinician on the basis of the physical health check and the available medical information.
* Presence of electronic or metallic implants contraindicated to MRI scanning at 3 Tesla, or presence of any other contraindication to MRI
* History of asthma
* History of epilepsy or any other seizure
* Under 18 years of age
* Lacking mental capacity to consent
* Current or previous use of NAC
* Currently prescribed clozapine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified:
  1. Via South London and Maudsley (SLaM) clinical teams.
  2. If they have previously indicated to local research teams that they would like to be contacted about future research.
  2. Through the SLaM NIHR Bioresource, including patients in CRIS, the research informatics database, who have given consent to be contacted about research projects.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-06; Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Reduction in brain glutamate | One hour post capsule
  The within-subjects difference in brain glutamate concentration following a single oral administration of placebo compared to 2400mg N-acetylcysteine

SECONDARY OUTCOMES:
Brain perfusion | One hour post capsule
  The within-subjects change in regional brain perfusion, as assessed using pulsed continuous arterial spin labelling (pCASL) MRI, following a single oral administration of placebo compared to 2400mg N-acetylcysteine.
Regional activity and connectivity | One hour post capsule
  The within-subjects change in regional brain activity or connectivity, as assessed using resting state functional magnetic resonance imaging (rsfMRI), following a single oral administration of placebo compared to 2400mg N-acetylcysteine.

CONTACTS AND LOCATIONS:
Overall Officials: James H McCabe, Principal Investigator — King's College London
Locations (1):
- Institute of Psychiatry, Psychology and Neuroscience, Denmark Hill, London, United Kingdom

REFERENCES:
- [Background] Egerton A, Brugger S, Raffin M, Barker GJ, Lythgoe DJ, McGuire PK, Stone JM. Anterior cingulate glutamate levels related to clinical status following treatment in first-episode schizophrenia. Neuropsychopharmacology. 2012 Oct;37(11):2515-21. doi: 10.1038/npp.2012.113. Epub 2012 Jul 4. PMID 22763619
- [Background] Demjaha A, Egerton A, Murray RM, Kapur S, Howes OD, Stone JM, McGuire PK. Antipsychotic treatment resistance in schizophrenia associated with elevated glutamate levels but normal dopamine function. Biol Psychiatry. 2014 Mar 1;75(5):e11-3. doi: 10.1016/j.biopsych.2013.06.011. Epub 2013 Jul 25. No abstract available. PMID 23890739
- [Background] Berk M, Copolov D, Dean O, Lu K, Jeavons S, Schapkaitz I, Anderson-Hunt M, Judd F, Katz F, Katz P, Ording-Jespersen S, Little J, Conus P, Cuenod M, Do KQ, Bush AI. N-acetyl cysteine as a glutathione precursor for schizophrenia--a double-blind, randomized, placebo-controlled trial. Biol Psychiatry. 2008 Sep 1;64(5):361-8. doi: 10.1016/j.biopsych.2008.03.004. Epub 2008 Apr 23. PMID 18436195